CLINICAL TRIAL: NCT02295072
Title: ActiveBrains: Effects of an Exercise-based Randomized Controlled Trial on Cognition, Brain Structure and Brain Function in Overweight/Obese Preadolescent Children
Brief Title: Effects of an Exercise Program on Cognition and Brain in Overweight/Obese Preadolescent Children
Acronym: ActiveBrains
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Collaborators: Centro de Investigación Biomédica (Unknown); Hospital Clinico Universitario San Cecilio (Other); Instituto Mixto Universitario Deporte y Salud (Unknown); Centro de Investigación Mente, Cerebro y Comportamiento (Unknown)
Responsible Party: Principal Investigator, Francisco B. Ortega Porcel, Ramón & Cajal Researcher Fellow. Doctor in Exercise Physiology from University of Granada and Doctor in Medical Science from Karolinska Institutet of Stockholm., Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DEP2013-47540-R
Record Dates: First submitted 2014-11-14; First posted 2014-11-20 (Estimated); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Cognitive Function 1, Social; Mental Health Wellness 1; Obesity; Overweight
Keywords: Exercise-based Randomized Controlled Trial; Brain structure; Brain function; Cognitive function; Physical fitness; Body Mass Index; Cardiovascular disease risk factors; Mental health; Stress; Neurology; Obesity; brain; risk factors; bone; bones; body composition
MeSH Terms: conditions — Obesity; Overweight; Psychological Well-Being

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): 2 Usual Physical Education sessions/week
- Intervention Group (Experimental): A 5-months physical exercise-based program (3-5 Physical Education after school sessions/week + 2 Usual Physical Education sessions/week)
  Interventions: Behavioral: A 5-months physical exercise-based program

INTERVENTIONS:
Behavioral: A 5-months physical exercise-based program — The physical exercise program consists of 3-5 after-school sessions/week of 90 min plus "exercise homework" in the weekends, and will focus on high-intensity aerobic exercise mainly.
  Arms: Intervention Group

SUMMARY:
The ActiveBrains project aims to examine whether a 5-months physical exercise program has benefits on cognition and brain, as well as on selected physical and mental health outcomes in preadolescent overweight/obese children.

DETAILED DESCRIPTION:
New advances in neuroelectric and neuroimaging technologies in the last years provide a golden opportunity to further explore and understand how cognition and brain function can be stimulated by environmental factors, such as exercise, and particularly to study whether physical activity influences brain development in early ages. The present study, namely the ActiveBrains project, aims to examine the effects of a 5-months physical exercise program on cognition and brain, as well as on selected physical and mental health outcomes in preadolescents overweight/obese children.

A total of 100 overweight/obese preadolescent children aged 9 to 10 years will be randomized into an exercise group (N=50) and a control group (N=50). For practical and feasibility reasons, the study will be conducted in 2 waves, a 1st wave with a sample of 30 and a 2nd wave with a sample of 75. In this regard, 15 children will be intervened within one academic year (5-month intervention) and 35 children will be intervened within the following academic year. The control group will receive the usual physical education sessions (2 per week). In order to study the extent to which the effect of the intervention remains or disappears once the formal intervention is finished, we will do a 3rd evaluation in a subsample (50 participants from the 1st wave) 9 months after the intervention has finished. Waitlist control group strategy will be used, through which the control group will also receive an after-school exercise program but later, after all the assessments of the effectiveness of the program have been completed.

Based on existing literature, we believe that a 5-months physical exercise program is potentially beneficial for the cognition and brain, and for the physical and mental health of the overweight/obese children participating.

ELIGIBILITY:
Inclusion Criteria:

* Preadolescent children of Tanner stage of I, II or III.
* Children of 8 to 11 years-old,
* Overweight or obese defined based on the sex-and-age specific body mass index standards of Cole (2002).
* Girls must not have menstruation.

Exclusion Criteria:

* Children with Attention-Deficit Hyperactivity Disorder or any other psychiatric disorder.
* Left-handed children.
* Children with medical problem that prevent to practice physical activity.

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Actual)
Dates: Start 2014-12; Primary Completion 2017-03 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Changes in Brain function and structure using magnetic resonance imaging (MRI) | 20 days during baselines and Post-evaluations (after intervention).
  10-15 mins of high resolution scanning, 10 mins of resting state and 20 mins of Diffusion Tensor Imaging
Brain and cognitive functioning assessment by electroencephalogram (EEG) | 20 days during baselines and Post-evaluations (after intervention).
  Assessment of the processing information and speed trought event-related brain potentials, cognitive function using a EEG and doing two cognitive tasks of attention and working memory.
Cognitive performance (DKEFS test battery) | 20 days during baselines and Post-evaluations (after intervention).
  Executive function assessment with a set of tests of the DKEFS test battery that provide an assessment of verbal and non-verbal intelligence, one's initiation of problem-solving behavior, fluency in generating visual patterns, creativity in drawing new designs, simultaneous processing in drawing the designs while observing the rules and restrictions of the task, and inhibiting previously drawn responses, spatial planning, rule learning, inhibition of impulsive and perseverative responding, cognitive inhibition, flexibility of thinking on a visual-motor sequencing task and relational memory
Academic achievement | 20 days during baselines and Post-evaluations (after intervention).
  Academic achievement is assessed using final school recorded scores and the III Woodcock-Muñoz Battery which includes 5 reading tests, 4 oral tests, 4 mathematics tests, 4 written language tests and 4 tests of academic language.

SECONDARY OUTCOMES:
Physical Fitness | 20 days during baselines and Post-evaluations (after intervention).
  Aerobic fitness, muscular strength and speed-agility, following the ALPHA fitness test battery. In addition aerobic fitness will be additionally assessed using a gas analyzer (General Electric Corporation) while performing and maximal incremental treadmill test modified for poorly fit children
Mental Health | 20 days during baselines and Post-evaluations (after intervention).
  Chronic Stress indicators and behaviour and personality tests.
Body fatness and bone mass | 20 days during baselines and Post-evaluations (after intervention).
  Body fatness and bone mass assessment using dual-energy X-ray absorciometry (DXA, Discovery densitometer from Hologic), following protocols used in previous studies
Cardio-metabolic risk factors | 20 days during baselines and Post-evaluations (after intervention).
  Here we will include a complete set of risk factors as markers of lipid profile (triglycerides and total-, HDL and LDL-cholesterol), blood pressure (following standard procedures), and insulin resistance (glucose and insulin, homeostasis model assessment, HOMA)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Cadenas-Sanchez C, Mora-Gonzalez J, Migueles JH, Martin-Matillas M, Gomez-Vida J, Escolano-Margarit MV, Maldonado J, Enriquez GM, Pastor-Villaescusa B, de Teresa C, Navarrete S, Lozano RM, de Dios Beas-Jimenez J, Estevez-Lopez F, Mena-Molina A, Heras MJ, Chillon P, Campoy C, Munoz-Hernandez V, Martinez-Avila WD, Merchan ME, Perales JC, Gil A, Verdejo-Garcia A, Aguilera CM, Ruiz JR, Labayen I, Catena A, Ortega FB. An exercise-based randomized controlled trial on brain, cognition, physical health and mental health in overweight/obese children (ActiveBrains project): Rationale, design and methods. Contemp Clin Trials. 2016 Mar;47:315-24. doi: 10.1016/j.cct.2016.02.007. Epub 2016 Feb 23. PMID 26924671
- [Result] Esteban-Cornejo I, Cadenas-Sanchez C, Contreras-Rodriguez O, Verdejo-Roman J, Mora-Gonzalez J, Migueles JH, Henriksson P, Davis CL, Verdejo-Garcia A, Catena A, Ortega FB. A whole brain volumetric approach in overweight/obese children: Examining the association with different physical fitness components and academic performance. The ActiveBrains project. Neuroimage. 2017 Oct 1;159:346-354. doi: 10.1016/j.neuroimage.2017.08.011. Epub 2017 Aug 5. PMID 28789992
- [Result] Rodriguez-Ayllon M, Cadenas-Sanchez C, Esteban-Cornejo I, Migueles JH, Mora-Gonzalez J, Henriksson P, Martin-Matillas M, Mena-Molina A, Molina-Garcia P, Estevez-Lopez F, Enriquez GM, Perales JC, Ruiz JR, Catena A, Ortega FB. Physical fitness and psychological health in overweight/obese children: A cross-sectional study from the ActiveBrains project. J Sci Med Sport. 2018 Feb;21(2):179-184. doi: 10.1016/j.jsams.2017.09.019. Epub 2017 Oct 4. PMID 29031643
- [Result] Esteban-Cornejo I, Rodriguez-Ayllon M, Verdejo-Roman J, Cadenas-Sanchez C, Mora-Gonzalez J, Chaddock-Heyman L, Raine LB, Stillman CM, Kramer AF, Erickson KI, Catena A, Ortega FB, Hillman CH. Physical Fitness, White Matter Volume and Academic Performance in Children: Findings From the ActiveBrains and FITKids2 Projects. Front Psychol. 2019 Feb 12;10:208. doi: 10.3389/fpsyg.2019.00208. eCollection 2019. PMID 30809168
- [Result] Plaza-Florido A, Migueles JH, Mora-Gonzalez J, Molina-Garcia P, Rodriguez-Ayllon M, Cadenas-Sanchez C, Esteban-Cornejo I, Solis-Urra P, de Teresa C, Gutierrez A, Michels N, Sacha J, Ortega FB. Heart Rate Is a Better Predictor of Cardiorespiratory Fitness Than Heart Rate Variability in Overweight/Obese Children: The ActiveBrains Project. Front Physiol. 2019 May 7;10:510. doi: 10.3389/fphys.2019.00510. eCollection 2019. PMID 31133870
- [Result] Adelantado-Renau M, Esteban-Cornejo I, Rodriguez-Ayllon M, Cadenas-Sanchez C, Gil-Cosano JJ, Mora-Gonzalez J, Solis-Urra P, Verdejo-Roman J, Aguilera CM, Escolano-Margarit MV, Verdejo-Garcia A, Catena A, Moliner-Urdiales D, Ortega FB. Inflammatory biomarkers and brain health indicators in children with overweight and obesity: The ActiveBrains project. Brain Behav Immun. 2019 Oct;81:588-597. doi: 10.1016/j.bbi.2019.07.020. Epub 2019 Jul 19. PMID 31330300
- [Result] Plaza-Florido A, Migueles JH, Mora-Gonzalez J, Molina-Garcia P, Rodriguez-Ayllon M, Cadenas-Sanchez C, Esteban-Cornejo I, Navarrete S, Maria Lozano R, Michels N, Sacha J, Ortega FB. The Role of Heart Rate on the Associations Between Body Composition and Heart Rate Variability in Children With Overweight/Obesity: The ActiveBrains Project. Front Physiol. 2019 Jul 16;10:895. doi: 10.3389/fphys.2019.00895. eCollection 2019. PMID 31379602
- [Result] Solis-Urra P, Esteban-Cornejo I, Cadenas-Sanchez C, Rodriguez-Ayllon M, Mora-Gonzalez J, Migueles JH, Labayen I, Verdejo-Roman J, Kramer AF, Erickson KI, Hillman CH, Catena A, Ortega FB. Early life factors, gray matter brain volume and academic performance in overweight/obese children: The ActiveBrains project. Neuroimage. 2019 Nov 15;202:116130. doi: 10.1016/j.neuroimage.2019.116130. Epub 2019 Aug 26. PMID 31465844
- [Result] Leppanen MH, Migueles JH, Cadenas-Sanchez C, Henriksson P, Mora-Gonzalez J, Henriksson H, Labayen I, Lof M, Esteban-Cornejo I, Ortega FB. Hip and wrist accelerometers showed consistent associations with fitness and fatness in children aged 8-12 years. Acta Paediatr. 2020 May;109(5):995-1003. doi: 10.1111/apa.15043. Epub 2019 Oct 20. PMID 31583747
- [Result] Ubago-Guisado E, Gracia-Marco L, Medrano M, Cadenas-Sanchez C, Arenaza L, Migueles JH, Mora-Gonzalez J, Tobalina I, Escolano-Margarit MV, Oses M, Martin-Matillas M, Labayen I, Ortega FB. Differences in areal bone mineral density between metabolically healthy and unhealthy overweight/obese children: the role of physical activity and cardiorespiratory fitness. Pediatr Res. 2020 Jun;87(7):1219-1225. doi: 10.1038/s41390-019-0708-x. Epub 2019 Dec 10. PMID 31822016
- [Result] Rodriguez-Ayllon M, Esteban-Cornejo I, Verdejo-Roman J, Muetzel RL, Migueles JH, Mora-Gonzalez J, Solis-Urra P, Erickson KI, Hillman CH, Catena A, Tiemeier H, Ortega FB. Physical Activity, Sedentary Behavior, and White Matter Microstructure in Children with Overweight or Obesity. Med Sci Sports Exerc. 2020 May;52(5):1218-1226. doi: 10.1249/MSS.0000000000002233. PMID 31876665
- [Result] Mora-Gonzalez J, Esteban-Cornejo I, Solis-Urra P, Migueles JH, Cadenas-Sanchez C, Molina-Garcia P, Rodriguez-Ayllon M, Hillman CH, Catena A, Pontifex MB, Ortega FB. Fitness, physical activity, sedentary time, inhibitory control, and neuroelectric activity in children with overweight or obesity: The ActiveBrains project. Psychophysiology. 2020 Jun;57(6):e13579. doi: 10.1111/psyp.13579. Epub 2020 Apr 6. PMID 32249933
- [Result] Zavala-Crichton JP, Esteban-Cornejo I, Solis-Urra P, Mora-Gonzalez J, Cadenas-Sanchez C, Rodriguez-Ayllon M, Migueles JH, Molina-Garcia P, Verdejo-Roman J, Kramer AF, Hillman CH, Erickson KI, Catena A, Ortega FB. Association of Sedentary Behavior with Brain Structure and Intelligence in Children with Overweight or Obesity: The ActiveBrains Project. J Clin Med. 2020 Apr 12;9(4):1101. doi: 10.3390/jcm9041101. PMID 32290576
- [Result] Rodriguez-Ayllon M, Esteban-Cornejo I, Verdejo-Roman J, Muetzel RL, Mora-Gonzalez J, Cadenas-Sanchez C, Plaza-Florido A, Molina-Garcia P, Kramer AF, Catena A, Ortega FB. Physical fitness and white matter microstructure in children with overweight or obesity: the ActiveBrains project. Sci Rep. 2020 Jul 27;10(1):12469. doi: 10.1038/s41598-020-67996-2. PMID 32719329
- [Result] Mora-Gonzalez J, Esteban-Cornejo I, Migueles JH, Rodriguez-Ayllon M, Molina-Garcia P, Cadenas-Sanchez C, Solis-Urra P, Plaza-Florido A, Kramer AF, Erickson KI, Hillman CH, Catena A, Ortega FB. Physical fitness and brain source localization during a working memory task in children with overweight/obesity: The ActiveBrains project. Dev Sci. 2021 May;24(3):e13048. doi: 10.1111/desc.13048. Epub 2020 Oct 25. PMID 33037758
- [Result] Esteban-Cornejo I, Stillman CM, Rodriguez-Ayllon M, Kramer AF, Hillman CH, Catena A, Erickson KI, Ortega FB. Physical fitness, hippocampal functional connectivity and academic performance in children with overweight/obesity: The ActiveBrains project. Brain Behav Immun. 2021 Jan;91:284-295. doi: 10.1016/j.bbi.2020.10.006. Epub 2020 Oct 10. PMID 33049365
- [Result] Plaza-Florido A, Altmae S, Esteban FJ, Cadenas-Sanchez C, Aguilera CM, Einarsdottir E, Katayama S, Krjutskov K, Kere J, Zaldivar F, Radom-Aizik S, Ortega FB. Distinct whole-blood transcriptome profile of children with metabolic healthy overweight/obesity compared to metabolic unhealthy overweight/obesity. Pediatr Res. 2021 May;89(7):1687-1694. doi: 10.1038/s41390-020-01276-7. Epub 2020 Nov 23. PMID 33230195
- [Derived] Gil-Cosano JJ, Ubago-Guisado E, Migueles JH, Cadenas-Sanchez C, Torres-Lopez LV, Martin-Matillas M, Labayen I, Ortega FB, Gracia-Marco L. A 20-week exercise program improved total body and legs bone mineral density in children with overweight or obesity: The ActiveBrains randomized controlled trial. J Sci Med Sport. 2024 Jan;27(1):3-9. doi: 10.1016/j.jsams.2023.10.005. Epub 2023 Oct 12. PMID 37891146
- [Derived] Migueles JH, Cadenas-Sanchez C, Lubans DR, Henriksson P, Torres-Lopez LV, Rodriguez-Ayllon M, Plaza-Florido A, Gil-Cosano JJ, Henriksson H, Escolano-Margarit MV, Gomez-Vida J, Maldonado J, Lof M, Ruiz JR, Labayen I, Ortega FB. Effects of an Exercise Program on Cardiometabolic and Mental Health in Children With Overweight or Obesity: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2023 Jul 3;6(7):e2324839. doi: 10.1001/jamanetworkopen.2023.24839. PMID 37498603
- [Derived] Ortega FB, Mora-Gonzalez J, Cadenas-Sanchez C, Esteban-Cornejo I, Migueles JH, Solis-Urra P, Verdejo-Roman J, Rodriguez-Ayllon M, Molina-Garcia P, Ruiz JR, Martinez-Vizcaino V, Hillman CH, Erickson KI, Kramer AF, Labayen I, Catena A. Effects of an Exercise Program on Brain Health Outcomes for Children With Overweight or Obesity: The ActiveBrains Randomized Clinical Trial. JAMA Netw Open. 2022 Aug 1;5(8):e2227893. doi: 10.1001/jamanetworkopen.2022.27893. PMID 36040742
- [Derived] Migueles JH, Cadenas-Sanchez C, Aguiar EJ, Molina-Garcia P, Solis-Urra P, Mora-Gonzalez J, Garcia-Marmol E, Shiroma EJ, Labayen I, Chillon P, Lof M, Tudor-Locke C, Ortega FB. Step-Based Metrics and Overall Physical Activity in Children With Overweight or Obesity: Cross-Sectional Study. JMIR Mhealth Uhealth. 2020 Apr 28;8(4):e14841. doi: 10.2196/14841. PMID 32343251
- [Derived] Nystrom CD, Henriksson P, Martinez-Vizcaino V, Medrano M, Cadenas-Sanchez C, Arias-Palencia NM, Lof M, Ruiz JR, Labayen I, Sanchez-Lopez M, Ortega FB. Does Cardiorespiratory Fitness Attenuate the Adverse Effects of Severe/Morbid Obesity on Cardiometabolic Risk and Insulin Resistance in Children? A Pooled Analysis. Diabetes Care. 2017 Nov;40(11):1580-1587. doi: 10.2337/dc17-1334. Epub 2017 Sep 22. PMID 28939688
- See also: Pubmed link Methodological — https://pubmed.ncbi.nlm.nih.gov/26924671/

DOCUMENTS (1):
  • Statistical Analysis Plan (2021-06-19): https://cdn.clinicaltrials.gov/large-docs/72/NCT02295072/SAP_000.pdf